CLINICAL TRIAL: NCT06021392
Title: Comparative Study Between Wide Local Excision and Minimal Excision of Pilonidal Sinus
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Abanoub emad fayez (Other)
Responsible Party: Sponsor-Investigator, Abanoub emad fayez, Resident doctor in Assiut university hospitals, Assiut University
Organization: Assiut University (Other)
Other Study IDs: Techniques of PNS excision
Record Dates: First submitted 2023-08-28; First posted 2023-09-01 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-09

CONDITIONS: Pilonidal Sinus
MeSH Terms: conditions — Pilonidal Sinus

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Wide local excision of pilonidal sinus
  Interventions: Procedure: Z plasty and minimal excision of pilonidal sinus
- Minimal excision of pilonidal sinus
  Interventions: Procedure: Z plasty and minimal excision of pilonidal sinus

INTERVENTIONS:
Procedure: Z plasty and minimal excision of pilonidal sinus — The investigators will perform a " Z plasty " procedure and Minimal excision procedure for patients complaining of pilonidal sinus and the investigators will compare the outcomes and rate of recurrence of these two procedures

SUMMARY:
Comparative study between wide local excision and minimal excision of pilonidal sinus

DETAILED DESCRIPTION:
Pilonidal sinus (PNS) disease is distributed in young adults who are supposed to be healthy with maximum productivity. Wide local excision creates a tissue gap, while the concept of minimal excision preserves healthy tissues with minimal tissue gap.

Pilonidal disease is a frequent suppurative condition that occurs twice as often in men as in women, usually between the ages of 15 and 30. Pilonidal disease is located beneath the skin of the sacro-coccygeal region. It presents acutely as an abscess under tension while the chronic form gives rise to intermittent discharge from pilonidal sinus(es). Diagnosis is clinical and usually straightforward. In the large majority of cases, treatment is surgical but there is no consensus as to the 'ideal' technique. Acute abscess must be evacuated and an off-midline incision seems preferable. Excision is the standard definitive treatment but the choice of wide versus limited excision on the school of thought. Minimal excision or debridement of the sinus and/or cavity through a midline or a separate paramedian excision can also be performed, leaving the wounds open or closed. These methods are simple and cost-efficient, and associated with low pain, rapid healing, and a rapid return to normal activity. A disadvantage is the higher recurrence rate; however, these methods can be used repeatedly for recurrences. Although recurrence rates seem high at first glance, the procedures can be successfully repeated for recurrences, achieving healing rates of over 90% for 1-2 interventions. Future well-designed trials are necessary to aid patient selection.

ELIGIBILITY:
Inclusion Criteria:

* Patients complaining of primary PNS and Recurrent PNS following Minimal excision

Exclusion Criteria:

* Recurrent PNS following wide local excision

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy people of both genders with or without history of PNS procedures before
Sampling Method: Probability Sample
Enrollment: 2 (Estimated)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Rate of recurrence | In about 6 month follow up
  Showing each of both procedures efficacy in decreasing rate of recurrence of PNS